CLINICAL TRIAL: NCT03880500
Title: MRI-quantified Changes in Perfusion and Diffusion in Spinal Segments After High-Velocity, Low-Amplitude Spinal Manipulation: A Randomized Controlled Trial
Brief Title: Spinal Segment MRI Perfusion and Diffusion Response to Spinal Manipulation in Low Back Pain Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Balgrist University Hospital (Other)
Collaborators: Verein Pro Chiropraktik (Unknown); Balgrist Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BalgristUH
Record Dates: First submitted 2018-12-06; First posted 2019-03-19 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Pain, Back
MeSH Terms: conditions — Back Pain

STUDY DESIGN:
Intervention Model Description: 20 Controls, 50 Patients
Who Masked: Investigator, Outcomes Assessor
Masking Description: Blinding of Investigator to type of Intervention Blinding of Outcome assesors during follow-up.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient (Sham Comparator): 25 Patients will receive a spinal manipulative therapy Intervention, the other 25 Patients receive a sham Intervention.
  Interventions: Other: Spinal Manipulative Therapy
- Control (No Intervention): No intervention

INTERVENTIONS:
Other: Spinal Manipulative Therapy — The patient lies in sidelying position, with the hip of the upper leg flexed to 90° and the foot of the flexed leg hooked behind the popliteal space of the downside leg. The chiropractor faces the subject at a 45°-angle, fixates the flexed knee with his own knee/thigh. The fingers of the cephalic hand reach under the patient's upper arm to contact the upside lateral surface of the superior spinous process. The fingers of the caudal hand hook down-side aspect of the spinous process, the forearm contacts the patient's buttock and thigh. The cephalic hand thrusts lateromedially and caudocranially, from upside toward downside (push). The caudal hand thrusts lateromedially in the opposing direction, from downside toward upside (pull). SMT is repeated after the patient turns to left side lying.
  Other Names: SMT; Spinal Manipulative Intervention; Thrust Manipulation; High-velocity, low-amplitude thrust
  Arms: Patient

SUMMARY:
The main objective is to quantify changes in diffusion and perfusion in the intervertebral disc and adjacent spinal muscle tissue of a spinal segment receiving a spinal manipulative or control intervention using diffusion-weighted magnetic resonance Imaging (MRI) (DWI, used for quantifying diffusion) and intravoxel incoherent motion MRI (IVIM, used for quantifying perfusion).

Additional objectives are to test if clinical parameters such as pain and disability, radiological parameters, or pain-related inflammatory parameters in venous blood have predictive value in relation to these perfusion and diffusion effects, and if these effects correlate to clinical outcome.

An additional objective is to test the repeatability of IVIM-MRI in assessing perfusion changes in musculoskeletal tissue, and, as a positive control, assessing diurnal changes in perfusion and diffusion parameters in spinal tissue of healthy controls.

DETAILED DESCRIPTION:
Non-specific low back pain (LBP) is a very common condition in developed countries, with a point prevalence between 15% and 30% and a lifetime prevalence of about 70%. As a non-invasive treatment method, high-velocity, low-amplitude spinal manipulative therapy (SMT) is used in the conservative treatment of non-specific low back pain (LBP). Several studies suggest an association with favourable outcome. However, the overall effect size of clinical improvement following SMT remains modest. Most research on the effectiveness of SMT on back pain is conducted on patients suffering from "non-specific" LBP, the diagnosis of which is usually based upon the criterium that pain is not attributed to a recognizable pathology (e.g., infection, tumor, inflammatory diseases, fractures, disc herniations with nerve compression)8. In most of these studies, it is unclear whether patients' diagnoses were based upon more than history and clinical examination. The investigators argue that in the majority of cases, back pain labelled as non-specific might be more accurately labelled as non-specified and does have an attributable source and cause, whether one is able to recognize it or not. Therefore, if the diagnosis of non-specific LBP comprises heterogenic conditions, it is unlikely that patients will respond to one therapeutic modality equally.

Diffusion-weighted MR-imaging (DWI) is an application of magnetic resonance imaging that allows the measurement of water movement within and between tissues and is increasingly being used to study musculoskeletal physiology. Because DWI is sensitive even to small changes in fluid flow, it is potentially valuable in the study of the influence of therapeutic interventions such as manual therapy, exercise, and physical agents on musculoskeletal tissues. Studies using DWI have suggested that changes in diffusion within lumbar intervertebral discs occur in response to joint mobilization, prone press-ups, spinal traction and spinal manipulative therapy.

Intravoxel incoherent motion (IVIM) is a method proposed in 1988 by Le Bihan et al. which extracts microvascular blood flow information from diffusion-weighted imaging acquired at different b-values. It is used to generate separate images of diffusion and perfusion without requiring the injection of exogenous contrast agents. Originally developed in brain studies, it has been used in recent years to study perfusion in musculoskeletal tissue. There is a paucity of research addressing physiological events following a SMT intervention for patients with low back pain. A deeper understanding of local biomechanical and neurophysiological effects of SMT interventions might help refine its utilization and improve its effectiveness.

The purpose of this study is to quantify changes in diffusion and perfusion parameters within the intervertebral disc and paraspinal muscle tissue of a spinal segment receiving a spinal manipulative or sham intervention and to evaluate whether those changes differ in spinal segments with or without degenerative changes in 50 low-back-pain patients.

Additionally, it is of interest to determine the relationships between baseline parameters and changes in diffusion and perfusion as well as the degree of degenerative changes. Post-intervention changes in segmental spinal muscle perfusion will also be investigated. There will be a clinical follow-up immediately after the second MRI and at 1 week,4 and 12 weeks.

The repeatability and diurnal variation of IVIM imaging in quantifying perfusion in musculoskeletal tissues will be assessed by comparing perfusion parameters of 20 controls who will not receive any intervention. The investigators will perform a diffusion- and perfusion-weighted MRI at the beginning of the visit in the morning, which is repeated after approximately 20 minutes of rest (lying supine). Controls will present for an additional MRI approximately 10 hours later in the evening of the same day.

In participants consenting to venipuncture, approximately 8 ml of venous blood will be withdrawn using serum collection tubes, allowed to clot, and then centrifuged. The resulting serum supernatant is stored in aliquots at Balgrist Campus at -80°C. It will be analysed at the end of data collection for pro- and anti-inflammatory markers (e.g. C-reactive Protein, Interleukin 1-beta, Interleukin 6 and Tumor Necrosis Factor) in order to determine the relationship between inflammatory markers and degenerative changes, pain duration, and pain and disability outcomes.

ELIGIBILITY:
Inclusion criteria:

Patients:

1. Persons over 18 years and under 75 years of age with low back pain of any duration clinically not attributable to "red flags" (infection, trauma, fractures, inflammatory illnesses).
2. Source of LBP clinically at the L4/5 or L5/S1 segment.
3. Duration of LBP is longer than 4 weeks
4. Obtained informed consent.

Controls:

1. Persons over 18 years and under 75 years of age who have not suffered from low back pain in the last year and have never experienced low back pain for longer than 7 consecutive days.
2. Obtained informed consent.

Exclusion criteria:

Subjects are excluded from enrolment if they

1. have undergone prior spinal surgery
2. have undergone facet joint, epidural or periradicular injections in the last 6 months
3. had a spinal manipulative therapy intervention in the past 2 weeks
4. have spinal abnormalities (benign or malignant tumors, congenital abnormalities, isthmic spondylolisthesis)
5. have any contraindication to spinal manipulative interventions or are deemed unable to tolerate SMT to both body sides (e.g. pain attributable to above mentioned red flags, inability to perform side-lying without pain, radiculopathy with motor deficits <M4-, severe spinal canal stenosis)
6. have any contraindication to MRI (e.g. heart pacemaker, metallic foreign body or claustrophobia)
7. have started a new prescription medication targeting blood circulation within the last 3 months
8. are pregnant or nursing
9. Subjects are excluded from venipuncture if they are known to be HIV-positive or have Hepatitis A, B, or C or have another systemic infection (excludes subjects from venipuncture). No study specific testing for HIV or Hepatitis A, B or C is performed.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2019-03-06 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Apparent Diffusion Coefficient Change | Measured on day 1 during the study
  Computed on diffusion-weighted MRI, refers to the mean diffusion in a voxel (on MRI). Apparent diffusion coefficient (ADC) is measured in the intervertebral disc and adjacent spinal muscle tissue in patients before and after an SMT- or control intervention and in controls before and after 20 minutes of lying supine. The computed difference is the Apparent Diffusion Coefficient Change.
Capillary Perfusion Change | Measured on day 1 during the study
  Also called pseudodiffusion or D*. Measured on IVIM-MRI in square millimeters per second. Perfusion in capillaries in spinal muscle tissue is measured in patients before and after an SMT- or control intervention and in controls before and after 20 minutes of lying supine. The computed difference equals the Capillary Perfusion Change.
Diffusion Change | Measured on day 1 during the study
  Measured on diffusion-weighted MRI in square millimeters per second. Diffusion (D) in intra- and extracellular compartments in the intervertebral disc and adjacent spinal muscle tissue is measured in patients before and after an SMT- or control intervention and in controls before and after 20 minutes of lying supine. The computed difference is the Diffusion Change.

SECONDARY OUTCOMES:
Change in Apparent Diffusion Coefficient (Control) | Measured approximately 9 hours after the first MRI, during the study
  Measured on MRI. Secondary outcomes are the diurnal changes of the apparent diffusion coefficient in musculoskeletal tissue in controls approximately 9 hours after the first MRI.
Change in Capillary Perfusion (Control) | Measured approximately 9 hours after the first MRI, during the study
  Secondary outcomes are the diurnal changes of capillary perfusion in musculoskeletal tissue in controls approximately 9 hours after the first MRI.
Diffusion change | Measured approximately 9 hours after the first MRI, during the study
  Secondary outcomes are the diurnal changes of diffusion in the intervertebral disc and adjacent spinal muscle tissue in controls approximately 9 hours after the first MRI.

OTHER OUTCOMES:
Pfirrmann-Grade | Measured on day 1, during the study
  The severity of degenerative changes classified according to the Pfirrmann-grade on MRI.
  Grade I: disc is homogeneous with bright hyperintense white signal intensity and normal disc height.
  Grade II: disc is inhomogeneous, but keeping the hyperintense white signal. Nucleus and annulus are clearly differentiated, and a gray horizontal band could be present. Disc height is normal.
  Grade III: disc is inhomogeneous with an intermittent gray signal intensity. Distinction between nucleus and annulus is unclear. Disc height is normal or slightly decreased Grade IV: Disc is inhomogeneous with a hypointense dark gray signal intensity. There is no more distinction between the nucleus and annulus. Disc height is slightly or moderately decreased.
  Grade V: Disc is inhomogeneous with a hypointense black signal intensity. There is no more difference between the nucleus and annulus. The disc space is collapsed.
Weishaupt-Grade | Measured on day 1, during the study
  The severity of degenerative changes classified according to the Weishaupt-Classification on MRI.
  0 Normal facet joint space (2±4 mm width)
  1. Narrowing of the facet joint space (< 2 mm) and/or small osteophytes and/or mild hypertrophy of the articular process
  2. Narrowing of the facet joint space and/or moderate osteophytes and/or moderate hypertrophy of the articular process and/or mild subarticular bone erosions
  3. Narrowing of the facet joint space and/or large osteophytes and/or severe hypertrophy of the articular process and/or severe subarticular bone erosions and/or subchondral cysts
Inflammatory Parameters (interleukins) | Measured on day 1, during the study, and up to 12 months after
  The concentration of pro- and anti-inflammatory markers (Interleukin 1-beta, 4, 6, and 8) in the obtained blood samples.
Inflammatory Parameters (CRP) | Measured on day 1, during the study
  The concentration of CRP in the obtained blood samples.
Inflammatory Parameters (TNF-alpha) | Measured on day 1, during the study
  The concentration of TNF-Alpha in the obtained blood samples.
Disability Change | Disability change is assessed at 1 week, 1 month and 3 months follow-up
  Change in Oswestry disability Index. The questionnaire contains ten topics: intensity of pain, lifting, ability to care for oneself, ability to walk, ability to sit, sexual function, ability to stand, social life, sleep quality, and ability to travel. Each category consists of 6 statements describing different scenarios in the patient's life relating to the category. The patient checks the statement which most precisely resembles their situation. Each question is scored on a scale of 0-5 with the first statement being zero and indicating the least disability and the last statement is scored 5 indicating the most disability. The scores for all questions answered are added, then multiplied by two to obtain the index (range 0 to 100).
Pain Change: NRS | Pain change is assessed at 1 week, 1 month and 3 months follow-up
  Change in pain on the numerical Rating scale NRS (11-point Scale ranging from 0 (no pain) to 10 (most pain).
Treatment-related adverse events | Treatment-related adverse events are assessed at all time points during the study, starting from the time of inclusion to completion of 3 months follow up
  Number of participants with treatment-related adverse events as defined in the study Protocol Chapter 8.2.4.

CONTACTS AND LOCATIONS:
Overall Officials: Petra Schweinhardt, PhD, MD, Principal Investigator — Balgrist University Hospital
Locations (1):
- University Hospital Balgrist, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Beattie PF, Butts R, Donley JW, Liuzzo DM. The within-session change in low back pain intensity following spinal manipulative therapy is related to differences in diffusion of water in the intervertebral discs of the upper lumbar spine and L5-S1. J Orthop Sports Phys Ther. 2014 Jan;44(1):19-29. doi: 10.2519/jospt.2014.4967. Epub 2013 Nov 21. PMID 24261925
- [Background] Le Bihan D. What can we see with IVIM MRI? Neuroimage. 2019 Feb 15;187:56-67. doi: 10.1016/j.neuroimage.2017.12.062. Epub 2017 Dec 22. PMID 29277647
- [Background] Nguyen A, Ledoux JB, Omoumi P, Becce F, Forget J, Federau C. Application of intravoxel incoherent motion perfusion imaging to shoulder muscles after a lift-off test of varying duration. NMR Biomed. 2016 Jan;29(1):66-73. doi: 10.1002/nbm.3449. PMID 26684052
- [Background] Wong AY, Parent EC, Dhillon SS, Prasad N, Kawchuk GN. Do participants with low back pain who respond to spinal manipulative therapy differ biomechanically from nonresponders, untreated controls or asymptomatic controls? Spine (Phila Pa 1976). 2015 Sep 1;40(17):1329-37. doi: 10.1097/BRS.0000000000000981. PMID 26020851
- [Background] Klyne DM, Barbe MF, Hodges PW. Systemic inflammatory profiles and their relationships with demographic, behavioural and clinical features in acute low back pain. Brain Behav Immun. 2017 Feb;60:84-92. doi: 10.1016/j.bbi.2016.10.003. Epub 2016 Oct 6. PMID 27720935
- [Background] Chou R, Huffman LH; American Pain Society; American College of Physicians. Nonpharmacologic therapies for acute and chronic low back pain: a review of the evidence for an American Pain Society/American College of Physicians clinical practice guideline. Ann Intern Med. 2007 Oct 2;147(7):492-504. doi: 10.7326/0003-4819-147-7-200710020-00007. PMID 17909210

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-22): https://cdn.clinicaltrials.gov/large-docs/00/NCT03880500/Prot_SAP_000.pdf